CLINICAL TRIAL: NCT06383416
Title: Incidence of Headache and Its Effect on Quality of Life in Geriatric Patients With Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer of internal physical therapy, Ahram Canadian University
Other Study IDs: P.T-INT-10/2023-522
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Geriatric Patients With Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neck pain by VAS — chronic neck pain will be assessed by visual analogue scale. Patients will fill out quality of life questionnaire and headache disability index.
  Other Names: headache disability index; SF-36 quality of life questionnaire

SUMMARY:
cross sectional study to detect the incidence of headache and its effect on quality of life in geriatric patients with chronic neck pain. Patients will fill out quality of life questionnaire and headache disability index. We will take information from the patients about:

* The frequency of headache occurrence.
* Visual analogue scale of chronic neck pain. Main measures: chronic neck pain will be assessed by visual analogue scale. Patients will fill out quality of life questionnaire and headache disability index.

ELIGIBILITY:
Inclusion Criteria:

- geriatric patient with neck pain from 1moth ago

Exclusion Criteria:

* patient with the following conditions autoimmune disease neurological disease have previous cervical surgery

Ages: 60 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: geriatric patients with age range from 60-70 suffering from neck pain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | one time
headache disability index | one time
SF-36 quality of life questionare | one time

CONTACTS AND LOCATIONS:
Locations (1):
- Ababa physical therapy center, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No